CLINICAL TRIAL: NCT06394440
Title: Clinical Evaluation of Self-Adhesive Bulk-Fill Composite Versus Conventional Nano-hybrid Composite in Cervical Cavities - A Randomized Controlled Clinical Trial
Brief Title: Clinical Evaluation of Self-Adhesive Bulk-Fill Composite Versus Conventional Nano-hybrid Composite in Cervical Cavities
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Misr International University (Other)
Responsible Party: Principal Investigator, Riham Kamal ElDessouky ElShazly, Teaching Assistant, Misr International University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MIU-IRB-2223-177
Record Dates: First submitted 2022-11-23; First posted 2024-05-01 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Cervical Caries
MeSH Terms: conditions — Root Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Self-Adhesive Bulkfill Composite Restoration (Experimental): Surefil One from Dentsply will be applied to one side of teeth that contain cervical cavities.
  Interventions: Combination Product: Self-Adhesive Bulkfill Composite (Surefil One)
- Nano-hybrid Composite (Active Comparator): Neospectra from Dentsply will be added after etching & bonding to the other side of the teeth that contain cervical cavities.
  Interventions: Combination Product: Self-Adhesive Bulkfill Composite (Surefil One)

INTERVENTIONS:
Combination Product: Self-Adhesive Bulkfill Composite (Surefil One) — It is a new self-adhesive bulkfill composite that requires no previous adhesive steps.

SUMMARY:
The aim of this randomized clinical trial is to compare the six months clinical performance of the self-adhesive bulk-fill composite with the conventional nano-hybrid composite in the cervical lesions of teeth in the esthetic zone. In addition, to evaluate patient's satisfaction towards the self-adhesive bulk-fill material and its total operatory time.

DETAILED DESCRIPTION:
Patient Selection Patients will be randomly recruited from Dental Clinics at Misr International University (MIU) in Cairo. Written and signed informed consents will be obtained from all patients before participating in the clinical study after being completely informed of the aims, settings, procedures, benefits, and potential side effects of the study. The form will be approved by MIU's Ethical Committee. Patients will be selected according to the inclusion and exclusion criteria, carefully diagnosed, and will be allowed to read and understand the terms and conditions of the study and subsequently sign the informed consent. A total of 54 cervical lesions will be referred to be restored in this study. Materials will be randomly assigned to each side, considering that each patient must at least include two teeth and if more, even numbers of the cervical lesions will be selected. Patients will have all their selected teeth restored on their first visit. The randomization will be performed using Microsoft Excel (Microsoft, Washington, USA) by an independent contributor. Cervical lesions will be prepared, isolated and filled with the chosen material according to randomization.

Clinical Procedures The materials that will be used to restore cervical lesions in this study are self-adhesive bulk-fill composite (Surefil One, Dentsply Sirona) and Nanohybrid composite. Materials will be used according to manufacturer's instructions. Class V cavities will be prepared, restored, finished, and polished. Each patient will at least have one tooth restored by Surefil One and one tooth at least will be restored by conventional nano-hybrid composite.

For each patient, shade selection will be performed and accordingly the suitable shade of the composite will be selected before the start of any procedure using a dental shade guide. Local anesthesia will be given at the operation site and cervical cavities on the buccal surfaces will be prepared using 330 bur and finished using a red-coded stone to finish enamel margins and to create a bevel at the incisal margin of the cavity. Rubber dam will be placed on teeth restored to isolate the operative field before the initiation of the restorative process and a stopwatch will be used to record the time taken to place both restorations; starting from their application inside the cavity and the recording will be terminated right after finishing the restorative procedures.

Intervention At least one tooth in each patient will be restored with Surefil One capsule, following manufacturer's instructions, without any prior adhesive preparations. Capsule will be placed in the automatic mixer and mixed for six to eight seconds. Cleaning of the cavity will be achieved using an air-water spray leaving a moist cavity surface. The activated capsule will be attached to the applicator gun and the material is inserted inside the cavity at the deepest portion and gradually withdrawn allowing slight overfilling. Once the restorative material is applied and excess is removed using a hand instrument, restoration will be light cured using a LED Light Curing unit. The tip of the light unit will be put in contact with the glass slide during the light-curing process. The distance between the light source and the restoration will be standardized using a standard slide to ensure fixed curing distance. Rubber dam will be removed subsequently, and the finishing process of the material will be initiated using discs and finishing stones while the restoration is moist. A single step polishing protocol is followed consequently.

Comparator In the same patient, at least one tooth will be restored by conventional nano-hybrid composite. Etching of the enamel margins by 37% phosphoric acid will be done, rinsing with water after 20 seconds afterwards, drying using air blowing, followed by active application of two layers of Prime & Bond universal adhesive (Dentsply Sirona, Konstanz, Germany) using a micro-brush to the cavity, a waiting period of 15 seconds to allow the optimum penetration of the adhesive and curing for 20 seconds. Restorative material will be added incrementally, an increment of 2 mm thickness will be added, and light cured. Finishing of restorations will be done simultaneously after rubber dam removal using finishing discs and finishing stones. Restorations will be subsequently polished using a single step protocol of polishing.

Evaluation Procedures Cervical restorations will be inspected at baseline and after six months of restoration placement. The principal investigator will make sure to call each patient prior to their recall appointment to make sure that they show up exactly on the date and at the time of their follow up appointments. Restorations will be examined by two trained external blinded evaluators immediately after placing of restorations and their subsequent finishing and polishing without knowing which material was used in each cavity.

The USPHS criteria are selected and modified to suit the criteria chosen for the restoration evaluation. Evaluation instruments are dental mirrors, explorers, and intraoral photographs. Radiographs will only be taken if clinically indicated, for example caries diagnosis or pain experience. Adverse events regarding product safety will be recorded. Color match, surface roughness, marginal discoloration, marginal adaptation, retention, and the presence of secondary caries around restorations will be evaluated at baseline and after six months as a primary outcome. In addition, patient's satisfaction with the restoration will be measured immediately post-operative using Visual Analogue Scale (VAS) scores and the time elapsed from the start of isolation till finishing and polishing of the interventional restoration will be measured and compared to the time elapsed when restoring using a conventional composite. All observations will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Cervical lesions.
* Cervical lesions of at least one mm depth; to include enamel and dentin.
* Cervical lesions of not more than 3 mm in depth.
* Male or female genders.
* Medically free patients.
* Normal occlusion.
* Healthy Gingiva

Exclusion Criteria:

* Teeth showing signs of pulpitis or periapical pathosis.
* Patients older than 60 years.
* Patients younger than 18 years old.
* Pregnant women.
* Patients with history of allergy to resin.
* Patients with disabilities.
* Carious cervical lesions extending to proximal surfaces.
* Carious cervical lesions on the palatal/lingual surfaces.
* Teeth with root caries.
* Endodontically treated teeth.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-03-14 (Actual); Primary Completion 2024-07-20 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Clinical efficacy of the self-adhesive bulkfil composite in comparison to conventional composite | Six months
  Modified USPHS Criteria Alpha(A) Bravo(B) Charlie(C)

SECONDARY OUTCOMES:
Patient's Satisfaction of the final restorations | Six Months.
  Visual Analogue Scale (VAS). A scale 0-10; 0 - Extremely unsatisfactory 5 - Neutral 10 - Extremely satisfactory

CONTACTS AND LOCATIONS:
Locations (1):
- Misr International University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 5 Years
Access Criteria: Clinicaltrials.gov
URL: http://clinicaltrials.gov